CLINICAL TRIAL: NCT04288921
Title: A Multicenter Study Conducted to Evaluate the Performance of the LumiraDx Influenza A/B + RSV Test at Point of Care Testing Sites
Brief Title: Evaluation of Performance of the LumiraDx Influenza A/B + RSV Test at POC Testing Sites
Acronym: INSPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00015
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Influenza, Human; Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Influenza, Human; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: A performance evaluation study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Nasal swab (Experimental): Nasal swab from subjects with signs and symptoms of influenza and/or RSV-like illness
  Interventions: Diagnostic Test: Swab
- Nasopharyngeal swab (Experimental): Nasopharyngeal swab from subjects with signs and symptoms of influenza and/or RSV-like illness
  Interventions: Diagnostic Test: Swab

INTERVENTIONS:
Diagnostic Test: Swab — Swab samples for diagnostic test

SUMMARY:
A Multicenter Study Conducted to Evaluate the Performance of the LumiraDx Influenza A/B + RSV Test at Point of Care Testing Sites

DETAILED DESCRIPTION:
The LumiraDx Influenza A/B + RSV Test is a rapid microfluidic immunofluorescence assay for use with the LumiraDx instrument for the qualitative detection and differentiation of Influenza type A, Influenza type B and respiratory syncytial virus (RSV) viral antigens. The test is not intended to detect influenza C antigens. The LumiraDx Influenza A/B + RSV assay uses nasal swabs or nasopharyngeal swab specimens, collected from symptomatic patients.

Approximately 2000 subjects will be enrolled in this study. 120 influenza A positive, 120 influenza B positive and 120 RSV positive samples are required, in addition to at least 120 samples negative for influenza and 120 negative RSV samples, representing four (4) age groups: ≤ 5 years, 6 to 21 years, 22 to 59 years, and ≥ 60 years. Depending on the prevalence of influenza A, influenza B or RSV, it will be necessary to collect a significantly higher number of total samples to obtain the required number of positives. Banked specimens may be used to supplement the data set.

The objectives of this clinical study are twofold:

* Evaluate the performance of the LumiraDx Influenza A/B + RSV Test in detecting and differentiating influenza A, influenza B and RSV in fresh nasal or nasopharyngeal swab specimens from patients with signs and symptoms of influenza and or RSV-like illness, as compared with an FDA-cleared comparative method.
* Evaluate LumiraDx Influenza A/B + RSV Test performance when the test is run by non-laboratory users in point-of-care (POC) locations representative of sites who perform testing under a CLIA certificate of waiver.

ELIGIBILITY:
Inclusion Criteria:

* The subject may be of any age and either sex.
* Preliminary assessment of the subject by the Investigator/designee should be suggestive of influenza and/or RSV at the time of the study visit. The subject must exhibit two (2) or more of the following signs and symptoms for eligibility: stuffy or runny nose, sneezing, cough, sore throat, dyspnea (labored, difficult breathing), wheezing, fatigue, weakness and/or malaise, arthralgia (joint pain), myalgia (deep muscle aches), anorexia, vomiting, diarrhea, or headache. The onset of these symptoms must not have begun more than four (4) days prior to study enrollment.
* The subject must have a fever of 100.0 °F or greater with the onset of the fever being within the past three (3) days and/or present at the time of the visit. Fever can be reported or taken at time of visit. Subjects 18 years and older must report having a fever, but a quantitative reported measurement is not necessary for inclusion.

Exclusion Criteria:

* The subject underwent a nasal wash/aspirate as part of standard of care testing during this study visit.
* The subject is undergoing treatment currently and/or within the past 14 days of the study visit with an inhaled influenza vaccine (FluMist®) or anti-viral medication, which may include but is not limited to Amantadine (Symmetrel®), Rimantadine (Flumadine®), Zanamivir (Relenza®), Oseltamivir (Tamiflu®), or Baloxavir Marboxil (Xofluza™).
* The subject is undergoing treatment currently or had undergone within the past 14 days of the study visit with RSV-related medication which may include but is not limited to Ribavirin (Virazole), RSV-IGIV (RespiGam) or palivizumab (Synagis).
* The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
* The subject has previously participated in this research study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Performance evaluation by health care professionals | 4 months
  Evaluate the performance of the LumiraDx Influenza A/B + RSV Test in detecting and differentiating influenza A, influenza B and RSV in fresh nasal or nasopharyngeal swab specimens from patients with signs and symptoms of influenza and or RSV-like illness, as compared with an FDA-cleared comparative method.
Performance evaluation by non-laboratory users | 4 months
  Evaluate LumiraDx Influenza A/B + RSV Test performance when the test is run by non-laboratory users in point-of-care (POC) locations representative of sites who perform testing under a CLIA certificate of waiver.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Ulen, Principal Investigator — Advanced Pediatrics; Robert Rosen, Principal Investigator — Ardmore Family Practice; Ramin Farsad, Principal Investigator — Access Medical Center; Matthew Morgan, Principal Investigator — Centura Health Physician Group; Jeffrey Stewart, Principal Investigator — Family Medical Associates; Andre Gvozden, Principal Investigator — Gvozden Pediatrics; Isaac Melamed, Principal Investigator — ImmunoE Health Center; Nader Nakhleh, Principal Investigator — Jersey Shore UMC; Lisa Connery, Principal Investigator — Lisa Connery MD; Aftab Naz, Principal Investigator — Madera Family Medical Group; Salma Elfaki, Principal Investigator — Nona Pediatric Center; Adam Kaplan, Principal Investigator — North Texas Family Practice; Paul Wisman, Principal Investigator — Pediatric Research of Charlottesville; William Simon, Principal Investigator — New Medical Healthcare; Joshua Fuller, Principal Investigator — Pediatric Care; David King, Principal Investigator — Southwest Care; Song Yu, Principal Investigator — MedHelp Urgent Care; Michael Bell, Principal Investigator — Accel-West Volusia Pediatrics
Locations (20):
- United States (20):
  - MedHelp Urgent Care, Birmingham, Alabama
  - Access Medical Center, Encinitas, California
  - Madera Family Medical Group, Madera, California
  - ImmunoE Health and Research, Centennial, Colorado
  - Complete Family Care Research, Northglenn, Colorado
  - ImmunoE Health and Research Center, Thornton, Colorado
  - Accel-West Volusia Pediatrics, DeLand, Florida
  - Nona Pediatric Center, Orlando, Florida
  - New Medical, Wichita, Kansas
  - Gvozden Pediatrics, Millersville, Maryland
  - Kent Plaza Pediatrics, Jackson, New Jersey
  - Jersey Shore UMC, Neptune City, New Jersey
  - Southwest Care, Santa Fe, New Mexico
  - Ardmore Family Practice, Winston-Salem, North Carolina
  - Lisa Connery MD, Norman, Oklahoma
  - Family Medical Associates, Carrollton, Texas
  - North Texas Family Practice, Plano, Texas
  - Pediatric Care, Bountiful, Utah
  - Pediatric Associates of Charlottesville, Charlottesville, Virginia
  - Advanced Pediatrics, Vienna, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellis JE, Guest P, Lawson V, Loecherbach J, Lindner N, McCulloch A. Performance Evaluation of the Microfluidic Antigen LumiraDx SARS-CoV-2 and Flu A/B Test in Diagnosing COVID-19 and Influenza in Patients with Respiratory Symptoms. Infect Dis Ther. 2022 Dec;11(6):2099-2109. doi: 10.1007/s40121-022-00696-8. Epub 2022 Sep 24. PMID 36152227